CLINICAL TRIAL: NCT06212700
Title: Virtual Multimodal Hub for Patients Undergoing Major Gastrointestinal Cancer Surgery - PRIORITY-CONNECT 2 Pilot Randomised Type I Hybrid Effectiveness-Implementation Trial
Brief Title: PRIORITY-CONNECT 2 Pilot Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Surgical Outcomes Research Centre (SOuRCe) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: X23-0399
Record Dates: First submitted 2023-12-13; First posted 2024-01-19 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Liver Cancer; Pancreas Cancer; Oesophageal Cancer; Gastric Cancer; Colorectal Cancer
Keywords: Prehabilitation; Gastrointestinal cancer; Surgery; Surgical outcomes; Randomised controlled trial
MeSH Terms: conditions — Liver Neoplasms; Pancreatic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Colorectal Neoplasms; Gastrointestinal Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: Randomised Type I Hybrid Effectiveness-Implementation Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Consenting participants will undergo baseline assessment immediately prior to randomisation to intervention (virtual multimodal hub and usual care) or control group (usual care alone). The randomisation sequence will be prepared a priori using a central secure randomisation service (1:1 allocation ratio in random permuted blocks of sizes 4 or 2 stratified by hospital, to ensure balance intreatment assignment within hospital) to ensure concealment of treatment allocation and blinding of surgeon, all trial personnel and statistician. Due to the nature of the intervention, it is not possible to blind the clinicians delivering the intervention (virtual multimodal hub); however, the investigators will ensure that all patients' interactions are standardised.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Multimodal Hub and usual care (Intervention Group) (Experimental): The main aim of the virtual multimodal hub is to prepare participants for surgery (including the role of Enhanced Recovery after Surgery (ERAS) pathway) and support declines in physiological and psychological function associated with preoperative treatments (e.g., chemo-radiotherapy) and major surgery. The post-hospital discharge interventions will focus on the recovery of activities of daily living, occupational tasks, and recreational activities. Aided by standardised assessment tools, a comprehensive holistic baseline (first preoperative multimodal session) and post-discharge (first postoperative multimodal session) assessment of patients' physical, nutritional, psychological and overall health status, presence of co-morbidities and medical history will determine the frequency, intensity, time, type, volume, and progression of the multimodal interventions.
  Interventions: Behavioral: Preoperative Exercise; Behavioral: Postoperative Exercise; Dietary Supplement: Preoperative Nutrition; Dietary Supplement: Postoperative Nutrition; Behavioral: Preoperative Psychology; Behavioral: Postoperative Psychology; Other: Preoperative Nursing; Other: Postoperative Nursing; Other: Preoperative Peer Support Group; Other: Postoperative Peer Support Group; Other: Usual Care
- Usual care alone (Control Group) (Active Comparator): Participants allocated to the control group will receive usual care according to their health care team, which may consist of advice on smoking cessation, reduction of alcohol intake, nutritional counselling, and medical optimisation in the preoperative anaesthetic clinic visits. Participants will be asked to maintain their normal daily activities.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Preoperative Exercise — Aerobic (HIIT) Endurance Respiratory Muscle Strength Education
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Behavioral: Postoperative Exercise — Aerobic Muscle Strength Walking Program Education
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Dietary Supplement: Preoperative Nutrition — Malnutrition screening Weight monitoring Symptom management Dietetic counselling Nutrition support
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Dietary Supplement: Postoperative Nutrition — Malnutrition screening Weight monitoring Symptom management Dietetic counselling Nutrition support
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Behavioral: Preoperative Psychology — CBT skills Skills training Emotional validation Behavioural activation Psycho-education
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Behavioral: Postoperative Psychology — CBT skills Skills training Emotional validation Behavioural activation Psycho-education
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Other: Preoperative Nursing — Comorbidities Managing pain Wound care Complications Surgical education ERAS
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Other: Postoperative Nursing — Managing pain Cardiovascular stability Wound care Bowel function/Stoma Complications Education
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Other: Preoperative Peer Support Group — Weekly sessions moderated by a social worker including patients and carers:
  Safe space Share experiences/ideas Support Education
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Other: Postoperative Peer Support Group — Weekly sessions moderated by a social worker including patients and carers:
  Safe space Share experiences/ideas Support Education
  Arms: Virtual Multimodal Hub and usual care (Intervention Group)
Other: Usual Care — Participants allocated to the control group will receive usual care according to their health care team, which may consist of advice on smoking cessation, reduction of alcohol intake, nutritional counselling, and medical optimisation in the preoperative anaesthetic clinic visits.

SUMMARY:
The provision of preoperative interventions (prehabilitation: including exercise, nutrition, and psychological treatment) have been reported to reduce postoperative complications by as much as 50% and reduce hospital stay by up to 4 days compared to standard of care. Postoperative multimodal interventions are likely to further benefit patients facing new challenges (e.g. stoma care), and reduce post discharge complications.

Therefore the Virtual Multimodal hub of PRIORITY-CONNECT 2 Pilot Trial aims to primarily; determine the feasibility of incorporating a virtual multimodal program into the preoperative and postoperative period for patients undergoing gastrointestinal cancer surgery, the acceptability to patients, clinicians and carers of the virtual multimodal program and the acceptability to patients of being randomised to the virtual multimodal program or usual care.

The secondary aim is to obtain pilot data on the likely difference in key outcomes (30 days postoperative complications, quality of life, days at home and alive at 30 days - DAH30, implementation outcomes and cost outcomes) to inform the development of a substantive randomised clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years undergoing major gastrointestinal elective surgery, including liver, pancreas, oesophagus, gastric and colorectal cancer resections with curative intent
* Consulting with a gastrointestinal cancer surgeon at least 1 week prior to scheduled surgery

Exclusion Criteria:

* Cognitive impairment such that they are unable to provide informed consent
* No access to a smart device (including mobile phone, tablet, laptop or desk computer with camera) or no internet connection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-07-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the virtual multimodal hub determined by number of eligible participants, retention rate and adherence rates | through study completion, an average of 1 year
  Feasibility will be determined by the following outcomes:
  (i) Number of eligible participants recruited to the pilot trial; (ii) Retention rate: defined as the percentage of participants who completed the trial; (iii) Adherence rates: defined as the percentage of planned sessions attended by those who were randomised to the intervention group.
Acceptability of the virtual multimodal hub. | 3 months, through study completion, an average of 1 year
  Patients, clinicians and carers acceptability to the virtual multimodal hub (Intervention) will be assessed with a semi-structured questionnaire administered at 3-months (last survey). The semi- structured questionnaire contains 11 questions and participants (Patients, clinicians and carers) will be instructed to use a 5-point Likert Scale to express how much they agree or disagree with each statement. In addition, patients will be asked how satisfied they were with the virtual multimodal program and if the program negatively affected them. The investigators have also taken the opportunity to seek further feedback about the virtual multimodal hub (open ended question). The questionnaire has been used on previous pilot trials.

SECONDARY OUTCOMES:
Postoperative complications within 30 days after surgery | 30 days after surgery
  Defined as any deviation from the normal postoperative course and classified according to the Clavien-Dindo classification. The risk of developing complications following gastrointestinal cancer surgery is highest in the first 30-days after surgery; this is a critical determinant of recovery, long-term outcomes, and gastrointestinal cancer treatment costs.
Quality of life outcome EORTC QLQ-C30 | Measured at baseline, 1-2 day(s) before surgery, day of hospital discharge, 1- and 3-months post index surgery.
  EORTC QLQ-C30 (European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire) is a 30-item cancer-specific tool measuring five functioning scales, nine symptom scales, financial impact and overall QoL. This tool is a common (excellent reliability and validity) QoL tool for gastrointestinal cancer patients. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Quality of life outcome EORTC QLQ-OG25 | Measured at baseline, 1-2 day(s) before surgery, day of hospital discharge, 1- and 3-months post index surgery.
  EORTC QLQ-OG25 (European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire) is a 25-item tool measuring function and symptoms specific to oesophoago-gastric cancer. This tool is a common (excellent reliability and validity) QoL tool for gastrointestinal cancer patients. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Quality of life outcome EORTC QLQ-CR29 | Measured at baseline, 1-2 day(s) before surgery, day of hospital discharge, 1- and 3-months post index surgery.
  EORTC QLQ-CR29 (European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire) is a 29-item tool measuring function and symptoms specific to colorectal cancer. This tool is a common (excellent reliability and validity) QoL tool for gastrointestinal cancer patients. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Number of days at home within 30 and 90 days of surgery | days at home within 30 and 90 days of surgery
  DAH-30, 90 (days at home 30, 90): Validated (Australian population) patient-centred outcome metrics that integrates length of hospital stay, discharge destination (other than home), hospital readmission and early death. The number of days at home - reduced by complications, discharge to a care facility, re-admission, and death is quantified as the days alive and at home during the 30 days after surgery. DAH-30, 90 is calculated using mortality and hospitalisation data from the date of the index surgery (= Day 0).
Resource use | 1-6 weeks prior to surgery to 3 months post index surgery.
  (Costs): Patient and health system resource use, including the cost of the virtual multimodal hub interventions, hospitalisations, will be collected (surveys) from randomisation (1-6 weeks prior to surgery) to 3 months post index surgery.
Implementation Outcome: Reach | through study completion, an average of 1 year
  RE-AIM Framework, including:
  Reach: Measured through trial participation, baseline characteristics (referral pathways, age, postcode, marital, work status, and Culturally And Linguistically Diverse [CALD]) of all potential participants.
Implementation Outcome: Effectiveness | through study completion, an average of 1 year
  RE-AIM Framework, including:
  Effectiveness: Measured through clinical outcomes, healthcare utilisation, participant satisfaction.
Implementation Outcome: Adoption | through study completion, an average of 1 year
  RE-AIM Framework, including:
  Adoption: Measured through referral rates, enablers and barriers (surveys with patients, carers, surgeons, clinical and administrative staff post intervention).
Implementation Outcome: Implementation | through study completion, an average of 1 year
  RE-AIM Framework, including:
  Implementation: measured through; Individual level: Participant adherence to virtual. Centre level: Implementation process, concordance with intervention protocol.
Implementation Outcome: Maintenance | through study completion, an average of 1 year
  RE-AIM Framework, including:
  Maintenance: Measured through rates of referral over time of the study; stakeholder interviews regarding refinements and infrastructure needed to maintain and scale intervention beyond the project period.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Chris O'Brien Lifehouse, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Surgical Outcomes Research Centre (SOuRCe), Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: No